CLINICAL TRIAL: NCT06258174
Title: A Phase I, Open-Label, Randomized, 2-Way Crossover Study to Compare the PK of Pirtobrutinib (LOXO-305) Tablets
Brief Title: A Study of Two Different Formulations of Pirtobrutinib (LOXO-305) In Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-BTK-21050; J2N-OX-JZNV (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Healthy
MeSH Terms: interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 200 mg Pirtobrutinib (Sequence R/T) (Experimental): Period 1: Participants received a reference formulation (R) of oral pirtobrutinib 200 milligrams (mg) on day 1.
  Period 2: Participants received a test formulation (T) of oral pirtobrutinib 200 mg on day 8.
  There was a washout period of 7 days between the doses of pirtobrutinib.
  Interventions: Drug: Pirtobrutinib
- 200 mg Pirtobrutinib (Sequence T/R) (Experimental): Period 1: Participants received a test formulation (T) of oral pirtobrutinib 200 mg on day 1.
  Period 2: Participants received a reference formulation (R) of oral pirtobrutinib 200 mg on day 8.
  There was a washout period of 7 days between the doses of pirtobrutinib.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally.
  Other Names: LOXO-305; LY3527727

SUMMARY:
The main purpose of this study is to compare two different formulations (mixtures) of pirtobrutinib (LOXO-305) in healthy participants. This study will compare how much of each formulation gets into the blood stream and how long it takes the body to remove it. Information about any side effects that may occur will be collected. The study will last up to 65 days.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of non-childbearing potential.
* Within body mass index (BMI) range 18.0 to 32.0 kilograms per square meter (kg/m²).
* Participants will be in good general health, based on medical history, physical examination findings, vital signs, 12 lead electrocardiogram (ECG), or clinical laboratory tests, as determined by the Investigator (or designee).

Exclusion Criteria:

* History or presence of any of the following, deemed clinically significant by the Investigator (or designee), and/or Sponsor:

  1. liver disease
  2. pancreatitis
  3. peptic ulcer disease
  4. intestinal malabsorption
  5. cholecystectomy
  6. gastric reduction surgery
  7. history or presence of clinically significant cardiovascular disease.
* Participants with out-of-range, at-rest vital signs.
* Abnormal laboratory values determined to be clinically significant by the Investigator (or designee).
* Clinically significant abnormality, as determined by the Investigator (or designee), from physical examination.
* Participation in any other investigational study drug trial involving administration of any investigational drug in the past 30 days or 5 half-lives, whichever was longer, prior to Day 1.
* Use or intention to use any prescription or over-the-counter medications within 14 days prior to Day 1 and through end of trial.
* History or presence, upon clinical evaluation, of any illness that, in the opinion of the Investigator, would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results, or put the participant at undue risk.
* Donation of blood from 56 days prior to Screening, plasma or platelets from 4 weeks prior to Screening.
* Receipt of blood products within 2 months prior to Check-in (Day -1).
* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, biliary, renal, hematological, pulmonary, cardiovascular (including any prior history of cardiomyopathy or cardiac failure), gastrointestinal (GI), neurological, or psychiatric disorder (as determined by the Investigator), or cancer within the past 5 years (except localized basal cell, squamous, or in situ cancer of the skin).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Ward, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Labcorp Drug Development, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to 2 treatment sequences (R/T, T/R), with each sequence having 2 periods where participants were crossed over between the periods. A washout period of 7 days was maintained between doses of each treatment period.
Period: Period 1
Arm/Group | 200 mg Pirtobrutinib (Sequence R/T) | 200 mg Pirtobrutinib (Sequence T/R)
Started | 14 | 14
Received at Least 1 Dose of Study Drug | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Period 2
Arm/Group | 200 mg Pirtobrutinib (Sequence R/T) | 200 mg Pirtobrutinib (Sequence T/R)
Started | 14 | 14
Received at Least 1 Dose of Study Drug | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 200 mg Pirtobrutinib (Sequence R/T): Period 1: Participants received a reference formulation (R) of oral pirtobrutinib 200 mg on day 1.
  Period 2: Participants received a test formulation (T) of oral pirtobrutinib 200 mg on day 8.
  There was a washout period of 7 days between the doses of pirtobrutinib.
- Total: Total of all reporting groups
Arm/Group | 200 mg Pirtobrutinib (Sequence R/T) | 200 mg Pirtobrutinib (Sequence T/R) | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (6.860) | 33.5 (9.940) | 36.9 (9.050)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 6 | 8 | 14
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time 0 to 24 Hours Post-dose (AUC0-24) of Pirtobrutinib
Description: PK: AUC0-24 of Pirtobrutinib
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: All randomized participants who received a dose of pirtobrutinib, had at least 1 quantifiable plasma concentration, and for whom at least 1 PK parameter was computed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- 200 mg Pirtobrutinib (Reference Formulation): Participants from R/T and T/R randomized sequences who received reference formulation (R) of oral pirtobrutinib 200 mg.
- 200 mg Pirtobrutinib (Test Formulation): Participants from R/T and T/R randomized sequences who received test formulation (T) of oral pirtobrutinib 200 mg.
Arm/Group | 200 mg Pirtobrutinib (Reference Formulation) | 200 mg Pirtobrutinib (Test Formulation)
Number analyzed (Participants) | 28 | 28
hour*nanogram per milliliter (h*ng/mL) | 48800 (29.1) | 49700 (20.6)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) of Pirtobrutinib
Description: PK: AUC0-t of Pirtobrutinib
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | 200 mg Pirtobrutinib (Reference Formulation) | 200 mg Pirtobrutinib (Test Formulation)
Number analyzed (Participants) | 28 | 28
hour*nanogram per milliliter (h*ng/mL) | 81100 (36) | 83600 (24.7)

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC0-inf) of Pirtobrutinib
Description: PK: AUC0-inf of Pirtobrutinib
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | 200 mg Pirtobrutinib (Reference Formulation) | 200 mg Pirtobrutinib (Test Formulation)
Number analyzed (Participants) | 28 | 28
hour*nanogram per milliliter (h*ng/mL) | 82000 (35.5) | 84700 (24.4)

4. Primary Outcome: PK: Percentage Extrapolation for AUC0-inf (%AUCextrap) of Pirtobrutinib
Description: PK: %AUCextrap of Pirtobrutinib
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUCextrap
Arm/Group | 200 mg Pirtobrutinib (Reference Formulation) | 200 mg Pirtobrutinib (Test Formulation)
Number analyzed (Participants) | 28 | 28
percentage of AUCextrap | 1.01 (46.9) | 1.12 (36.7)

5. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) of Pirtobrutinib
Description: PK: CL/F of Pirtobrutinib
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | 200 mg Pirtobrutinib (Reference Formulation) | 200 mg Pirtobrutinib (Test Formulation)
Number analyzed (Participants) | 28 | 28
liter per hour (L/h) | 2.44 (35.5) | 2.36 (24.4)

6. Primary Outcome: PK: Apparent Plasma Terminal Elimination Half-life (t1/2) of Pirtobrutinib
Description: PK: t1/2 of Pirtobrutinib
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | 200 mg Pirtobrutinib (Reference Formulation) | 200 mg Pirtobrutinib (Test Formulation)
Number analyzed (Participants) | 28 | 28
hours | 18.9 (21.2) | 19 (20.3)

7. Primary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) of Pirtobrutinib
Description: PK: Cmax of Pirtobrutinib
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | 200 mg Pirtobrutinib (Reference Formulation) | 200 mg Pirtobrutinib (Test Formulation)
Number analyzed (Participants) | 28 | 28
nanogram per milliliter (ng/mL) | 3960 (23.3) | 3980 (24.2)

8. Primary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Pirtobrutinib
Description: PK: Tmax of Pirtobrutinib
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Measure: Median (Full Range); unit: hours
Arm/Group | 200 mg Pirtobrutinib (Reference Formulation) | 200 mg Pirtobrutinib (Test Formulation)
Number analyzed (Participants) | 28 | 28
hours | 2.50 [0.500 to 6] | 2.50 [0.750 to 6]

9. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (λZ) of Pirtobrutinib
Description: PK: λZ of Pirtobrutinib
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: as for outcome 1
Measure: Number; unit: 1/hour (1/h)
Arm/Group | 200 mg Pirtobrutinib (Reference Formulation) | 200 mg Pirtobrutinib (Test Formulation)
Number analyzed (Participants) | 28 | 28
1/hour (1/h)
  Subject 1 | 0.0487 | 0.0347
  Subject 2 | 0.0420 | 0.0374
  Subject 3 | 0.0549 | 0.0563
  Subject 4 | 0.0446 | 0.0386
  Subject 5 | 0.0406 | 0.0382
  Subject 6 | 0.0382 | 0.0389
  Subject 7 | 0.0355 | 0.0348
  Subject 8 | 0.0335 | 0.0341
  Subject 9 | 0.0414 | 0.0390
  Subject 10 | 0.0431 | 0.0437
  Subject 11 | 0.0358 | 0.0321
  Subject 12 | 0.0432 | 0.0427
  Subject 13 | 0.0324 | 0.0382
  Subject 14 | 0.0198 | 0.0179
  Subject 15 | 0.0409 | 0.0371
  Subject 16 | 0.0457 | 0.0451
  Subject 17 | 0.0279 | 0.0284
  Subject 18 | 0.0305 | 0.0299
  Subject 19 | 0.0407 | 0.0478
  Subject 20 | 0.0290 | 0.0350
  Subject 21 | 0.0293 | 0.0342
  Subject 22 | 0.0408 | 0.0403
  Subject 23 | 0.0340 | 0.0322
  Subject 24 | 0.0269 | 0.0299
  Subject 25 | 0.0372 | 0.0379
  Subject 26 | 0.0359 | 0.0396
  Subject 27 | 0.0370 | 0.0369
  Subject 28 | 0.0360 | 0.0368

10. Primary Outcome: PK: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of Pirtobrutinib
Description: PK: Vz/F of Pirtobrutinib
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | 200 mg Pirtobrutinib (Reference Formulation) | 200 mg Pirtobrutinib (Test Formulation)
Number analyzed (Participants) | 28 | 28
Liter (L) | 66.6 (36.7) | 64.9 (28.4)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (Up To Day 24)
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | 200 mg Pirtobrutinib (Reference Formulation) | 200 mg Pirtobrutinib (Test Formulation)
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 1/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 200 mg Pirtobrutinib (Reference Formulation) (N=28) | 200 mg Pirtobrutinib (Test Formulation) (N=28)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT06258174/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT06258174/SAP_001.pdf